CLINICAL TRIAL: NCT03074643
Title: Long-term Effects of Weight Loss and Supplemental Protein on Physical Function
Brief Title: Utilizing Protein During Weight Loss to Impact Physical Function
Acronym: UPLIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00038668; R01AG050656 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Weight Loss; Diet Modification; Aging; Weight Change, Body; Dietary Habits
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight Changes; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: All participants will undergo a 6-month weight loss intervention of caloric restriction and supervised exercise followed by 12 months of follow-up with randomization to one of three groups (n=75/group): 1) Lower protein / higher CHO diet for the 6-month weight loss phase only (RecProt); 2) Higher protein / lower CHO diet for the 6-month weight loss phase only (6-mo HiProt); or 3) Higher protein / lower CHO diet for the 6-month weight loss and 12-month follow-up phases (18-mo HiProt).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- RecProt (Placebo Comparator): Lower protein / higher CHO diet for the 6-month weight loss phase. Exercise intervention months 0-6. Weight loss intervention months 0-6. Carbohydrate supplement for months 0-6 (blinded). Follow-up months 7-18.
  Interventions: Behavioral: Weight loss intervention months 0-6; Behavioral: Exercise intervention months 0-6; Dietary Supplement: Carbohydrate supplement for months 0-6
- 6-mon HiProt (Active Comparator): Higher protein / lower CHO diet for the 6-month weight loss phase. Exercise intervention months 0-6. Weight loss intervention months 0-6. Protein supplement for months 0-6 (blinded). Follow-up months 7-18.
  Interventions: Behavioral: Weight loss intervention months 0-6; Behavioral: Exercise intervention months 0-6; Dietary Supplement: Protein supplement for months 0-6
- 18-mon HiProt (Active Comparator): Higher protein / lower CHO diet for the 6-month weight loss and 12-month follow-up phases.
  Exercise intervention months 0-6. Weight loss intervention months 0-6. Protein supplement for months 0-6 (blinded). Protein supplement for follow-up months 7-18.
  Interventions: Behavioral: Weight loss intervention months 0-6; Behavioral: Exercise intervention months 0-6; Dietary Supplement: Protein supplement for months 0-6; Dietary Supplement: Protein supplement for follow-up months 7-18

INTERVENTIONS:
Behavioral: Weight loss intervention months 0-6 — All participants will undergo a dietary weight loss intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. The weight loss intervention will incorporate nutrition education (via group and individual meetings with the study dietitian), self-monitoring skills, cognitive-behavioral strategies for promoting lifestyle behavior modifications, and planned meals. Behavioral and educational group and individual sessions will be held weekly in a 3:1 ratio (3 group and 1 individual session per month).
Behavioral: Exercise intervention months 0-6 — All participants will be expected to participate in a supervised, center-based exercise program involving moderate-intensity aerobic exercise (e.g., treadmill walking) 3 days/wk during the 6-month weight loss intervention in accordance with the American Heart Association and the American College of Sports Medicine physical activity recommendations for older adults.
Dietary Supplement: Carbohydrate supplement for months 0-6 — Participants in the lower protein / higher CHO diet group (RecProt) will be provided a carbohydrate supplement (~50 g of carbohydrate and 220 calories) to consume daily during the 6 month weight loss intervention.
  Arms: RecProt
Dietary Supplement: Protein supplement for months 0-6 — Participants in the higher protein / lower CHO diet groups (6-mon HiProt and 18-mon HiProt) will be provided a protein supplement (~50 g of protein and 220 calories) to consume daily during the 6 month weight loss intervention.
  Arms: 18-mon HiProt; 6-mon HiProt
Dietary Supplement: Protein supplement for follow-up months 7-18 — Participants in the higher protein / lower CHO diet (18-mon HiProt) will be provided a protein supplement (~50 g of protein and 220 calories) to consume daily during the 12-month follow-up.
  Arms: 18-mon HiProt

SUMMARY:
This study will evaluate the effects of diet composition (i.e., amount of protein and carbohydrate) during a 6-month weight loss intervention and 12-months of follow-up on physical function, muscle mass, and weight loss maintenance in obese older adults. Participants will receive either a protein or carbohydrate supplement along with a behavioral weight loss intervention.

DETAILED DESCRIPTION:
The study will use a 3-group design in 225 obese (BMI 27-45 kg/m2), older (65-85 years) men and women at risk for disability (eSPPB <2.5) who will undergo a 6-month weight loss intervention followed by a 12-month follow-up phase to test the overall hypothesis that a higher protein (1.2 g/kg body wt/d) / lower carbohydrate (CHO) diet during a 6-month weight loss intervention improves physical function compared with an isocaloric lower protein (the current Recommended Dietary Allowance (RDA), 0.8 g/kg body wt/d) / higher CHO diet, and whether continuing a higher protein / lower CHO diet for 12-months following weight loss will result in better maintenance of improved physical function. All participants will undergo a 6-month weight loss intervention involving caloric restriction and supervised exercise followed by 12 months of follow-up with randomization to one of three groups (n=75/group): 1) Lower protein / higher CHO diet for the 6-month weight loss phase only (RecProt); 2) Higher protein / lower CHO diet for the 6-month weight loss phase only (6-mo HiProt); or 3) Higher protein / lower CHO diet for the 6-month weight loss and 12-month follow-up phases (18-mo HiProt). Physical function (primary aim) will be assessed by the expanded Short Physical Performance Battery (primary outcome) and lower extremity muscle strength at baseline, 6-, 12- and 18-months. Weight loss maintenance and body composition (secondary aim) will be assessed by dual-energy X-ray absorptiometry (DXA) and computed tomography (CT) at baseline, 6- and 18-months. Bone mineral density (DXA) and cardiometabolic risk factors will also be measured at baseline, 6- and 18-months.

ELIGIBILITY:
Inclusion Criteria:

* 65-85 years
* BMI: 27-45 kg/m2
* No regular resistance training and/or aerobic exercise (>20 mins/d) for past 6 months
* eSPPB <2.5
* No contraindications for safe and optimal participation in exercise training
* Approved for participation by Medical Director (Dr. Lyles)
* Willing to provide informed consent
* Agree to all study procedures and assessments
* Willing to consume protein/CHO supplements for up to 18 months
* Able to provide own transportation to study visits and intervention sessions

Exclusion Criteria:

* Weight loss (≥5%) in past 6 months
* Dependent on cane or walker
* Cognitive impairment (MoCA score <22)
* Severe arthritis, or other musculoskeletal disorder
* Joint replacement or other orthopedic surgery in past 6 months
* Uncontrolled resting hypertension (>160/90 mmHg);
* Insulin-dependent or uncontrolled diabetes (HbA1c ≥8%)
* Current or recent past (within 1 year) severe symptomatic heart disease, uncontrolled angina, stroke, chronic respiratory disease requiring oxygen; uncontrolled endocrine/metabolic disease; neurological or hematological disease; cancer requiring treatment in past year, except non-melanoma skin cancers; liver or renal disease; or clinically evident edema
* Unstable, severe depression
* Serious conduction disorder, uncontrolled arrhythmia, or new Q waves or ST-segment depressions (>3 mm at rest or ≥2 mm with exercise)
* Abnormal kidney function (eGFR <30 based on serum creatinine, age, gender, and race)
* Anemia (Hb<13 g/dL in men; <12 g/dL in women)
* Drug abuse or excessive alcohol use (>7 drinks/week women; >14 drinks/week men)
* Use of any tobacco or nicotine products in the past year
* Osteoporosis (T-score < -2.5 on hip or spine scan)
* Regular use of growth/steroid hormones, sex steroids or corticosteroids, osteoporosis medication, or protein supplements
* Weight loss medications or procedures
* Current participation in another intervention study

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Houston, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Geriatric Research Center at Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 6-month HiProt: Higher protein / lower CHO diet for the 6-month weight loss phase. Exercise intervention months 0-6. Weight loss intervention months 0-6. Protein supplement for months 0-6 (blinded). Follow-up months 7-18.
  Weight loss intervention months 0-6: All participants will undergo a dietary weight loss intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. The weight loss intervention will incorporate nutrition education (via group and individual meetings with the study dietitian), self-monitoring skills, cognitive-behavioral strategies for promoting lifestyle behavior modifications, and planned meals. Behavioral and educational group and individual sessions will be held weekly in a 3:1 ratio (3 group and 1 individual session per month).
  Exercise intervention months 0-6: All participants will be expected to participate in a supervised, center-based exercise program involving moderate-intensity aerobic exercise (e.g., treadmill walking) 3 days/wk during the 6-month weight loss intervention in accordance with the American Heart Association (AHA) and the American College of Sports Medicine (ACSM) physical activity recommendations for older adults.
  Protein supplement for months 0-6: Participants in the 6-month higher protein / lower CHO diet groups will be provided a protein supplement (~50 g of protein and 220 calories) to consume daily during the 6 month weight loss intervention.
- 18-month HiProt: Higher protein / lower CHO diet for the 6-month weight loss and 12-month follow-up phases.
  Exercise intervention months 0-6. Weight loss intervention months 0-6. Protein supplement for months 0-6 (blinded). Protein supplement for follow-up months 7-18.
  Weight loss intervention months 0-6: All participants will undergo a dietary weight loss intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. The weight loss intervention will incorporate nutrition education (via group and individual meetings with the study dietitian), self-monitoring skills, cognitive-behavioral strategies for promoting lifestyle behavior modifications, and planned meals. Behavioral and educational group and individual sessions will be held weekly in a 3:1 ratio (3 group and 1 individual session per month).
  Exercise intervention months 0-6: All participants will be expected to participate in a supervised, center-based exercise program involving moderate-intensity aerobic exercise (e.g., treadmill walking) 3 days/wk during the 6-month weight loss intervention in accordance with the AHA and the ACSM physical activity recommendations for older adults.
  Protein supplement for months 0-18: Participants in the 18-month higher protein / lower CHO diet groups will be provided a protein supplement (~50 g of protein and 220 calories) to consume daily during the 6 month weight loss intervention and 12 month follow-up.
Period: Overall Study
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt
Started | 62 | 62 | 63
Completed | 51 | 50 | 52
Not Completed | 11 | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt | Total
Number analyzed (Participants) | 62 | 62 | 63 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (4.4) | 71.8 (4.5) | 70.5 (3.9) | 71.0 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 42 | 124
  Male | 21 | 21 | 21 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 61 | 62 | 63 | 186
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 14 | 19 | 45
  White | 48 | 47 | 43 | 138
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body mass index (BMI) [Mean (Standard Deviation); unit: kg per meters squared] | 33.8 (4.6) | 34.3 (3.5) | 34.3 (4.2) | 34.2 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Expanded Short Physical Performance Battery Score
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet during a 6-month weight loss intervention and 12 months of follow-up on change in lower extremity physical function assessed by the expanded Short Physical Performance Battery score over 18 months. The expanded Short Physical Performance Battery score ranges from 0 to 4 with higher scores indicating better lower extremity physical function
Time Frame: 18 months
Population: 6 participants were missing the expanded Short Physical Performance battery at 18 month follow-up: 1 participant refused the test due to severe back pain (RecProt), 3 participants refused an in-person clinic visit due to COVID-19 concerns (1 per group); 1 participant moved out of state and only completed a phone visit (6-month HiProt); and 1 participant refused to complete the expanded Short Physical Performance Battery (6-month HiProt)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt
Number analyzed (Participants) | 49 | 47 | 51
score on a scale | 0.06 (0.08) | 0.11 (0.09) | 0.16 (0.09)
Statistical Analysis 1: Comparison: RecProt vs 18-month HiProt; Test type: Superiority; p = 0.16, ANCOVA; Adjusted for age, sex, race
Statistical Analysis 2: Comparison: 6-month HiProt vs 18-month HiProt; Test type: Superiority; p = 0.45, ANCOVA; Adjusted for age, sex, race

2. Secondary Outcome: Lower Extremity Muscle Strength
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet during a 6-month weight loss intervention and 12 months of follow-up on change in lower extremity muscle strength assessed using an isokinetic dynamometer (Biodex) over 18 months
Time Frame: 18 months
Population: 38 participants were missing leg strength: 34 were excluded from testing due to knee replacements, severe knee arthritis/pain, recent eye surgery or chest pain, history of brain aneurysms, or uncontrolled blood pressure (14 RecProt, 12 6-mo HiProt, 8 18-mo HiProt); 3 participants refused an in-person clinic visit due to COVID-19 concerns (1 per group); and 1 participant moved out of state and only completed a phone visit (6-mo HiProt)
Measure: Least Squares Mean (Standard Error); unit: Newton meters
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt
Number analyzed (Participants) | 36 | 36 | 43
Newton meters | 8.28 (4.81) | 6.27 (5.51) | 7.30 (5.27)
Statistical Analysis 1: Comparison: RecProt vs 18-month HiProt; Test type: Superiority; p = 0.81, ANCOVA; Adjusted for age, sex, race
Statistical Analysis 2: Comparison: 6-month HiProt vs 18-month HiProt; Test type: Superiority; p = 0.80, ANCOVA; Adjusted for age, sex, race

3. Secondary Outcome: Weight Change
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet during a 6-month weight loss intervention and 12 months of follow-up on change in body weight over 18 months
Time Frame: 18 months
Population: Weight was not available at 18 month follow-up in 2 participants: 1 participant moved out of state and only completed a phone visit (6-month HiProt) and 1 participant refused an in-person visit at 18 months due to COVID-19 concerns (RecProt)
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt
Number analyzed (Participants) | 50 | 49 | 52
kilograms | -2.67 (1.22) | -3.23 (1.26) | -3.28 (1.29)
Statistical Analysis 1: Comparison: RecProt vs 18-month HiProt; Test type: Superiority; p = 0.56, ANCOVA; Adjusted for age, sex, race
Statistical Analysis 2: Comparison: 6-month HiProt vs 18-month HiProt; Test type: Superiority; p = 0.96, ANCOVA; Adjusted for age, sex, race

4. Secondary Outcome: Total Body Lean Mass
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet during a 6-month weight loss intervention and 12 months of follow-up on change in dual energy x-ray (DXA) acquired total body lean mass over 18 months
Time Frame: 18 months
Population: 6 participants were missing DXA-acquired total body lean mass: 4 participants refused in-person visits due to COVID-19 concerns (1 RecProt, 1 6-m HiProt, 2 18-m HiProt), 1 participant moved out of state and only did a phone visit at follow-up (6-m HiProt), and there was a DXA machine malfunction for 1 participant (RecProt)
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt
Number analyzed (Participants) | 49 | 48 | 50
kilograms | -1.24 (0.48) | -1.68 (0.50) | -1.36 (0.52)
Statistical Analysis 1: Comparison: RecProt vs 18-month HiProt; Test type: Superiority; p = 0.76, ANCOVA; Adjusted for age, sex, race
Statistical Analysis 2: Comparison: 6-month HiProt vs 18-month HiProt; Test type: Superiority; p = 0.45, ANCOVA; Adjusted for age, sex, race

5. Secondary Outcome: Total Body Fat Mass
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet during a 6-month weight loss intervention and 12 months of follow-up on change in dual energy x-ray acquired (DXA) total body fat mass over 18 months
Time Frame: 18 months
Population: 6 participants were missing DXA-acquired total body fat mass: 4 participants refused in-person visits due to COVID-19 concerns (1 RecProt, 1 6-m HiProt, 2 18-m HiProt), 1 participant moved out of state and only did a phone visit at follow-up (6-m HiProt), and there was a DXA machine malfunction for 1 participant (RecProt)
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt
Number analyzed (Participants) | 49 | 48 | 50
kilograms | -1.47 (0.92) | -1.68 (0.95) | -1.72 (0.98)
Statistical Analysis 1: Comparison: RecProt vs 18-month HiProt; Test type: Superiority; p = 0.75, ANCOVA; Adjusted for age, sex, race
Statistical Analysis 2: Comparison: 6-month HiProt vs 18-month HiProt; Test type: Superiority; p = 0.95, ANCOVA; Adjusted for age, sex, race

6. Secondary Outcome: Thigh Muscle Volume
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet during a 6-month weight loss intervention and 12 months of follow-up on change in computerized tomography (CT) acquired thigh muscle volume over 18 months
Time Frame: 18 months
Population: 19 participants were missing CT-acquired thigh muscle volume: 10 participants refused the CT scan (5 RecProt, 2 6-m HiProt, 3 18-m HiProt); 4 participants had CT scans that were unable to be processed (1 RecProt, 1 6-m HiProt, 2 18-m HiProt); 3 participants refused in-person visits due to COVID-19 concerns (1 per group), 1 participant moved out of state and only did a phone visit at follow-up (6-m HiProt), and 1 person had a hip replacement of the leg scanned at baseline (18-m HiProt)
Measure: Least Squares Mean (Standard Error); unit: cm^3
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt
Number analyzed (Participants) | 44 | 45 | 45
cm^3 | -3.76 (2.77) | -5.40 (2.86) | -8.42 (2.96)
Statistical Analysis 1: Comparison: RecProt vs 18-month HiProt; Test type: Superiority; p = 0.06, ANCOVA; Adjusted for age, sex, race
Statistical Analysis 2: Comparison: 6-month HiProt vs 18-month HiProt; Test type: Superiority; p = 0.22, ANCOVA; Adjusted for age, sex, race

7. Secondary Outcome: Intermuscular Adipose Tissue
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet during a 6-month weight loss intervention and 12 months of follow-up on change in computerized tomography (CT) acquired thigh intermuscular adipose tissue over 18 months
Time Frame: 18 months
Population: 19 participants were missing CT-acquired intermuscular adipose tissue: 10 participants refused the CT scan (5 RecProt, 2 6-m HiProt, 3 18-m HiProt); 4 participants had CT scans that were unable to be processed (1 RecProt, 1 6-m HiProt, 2 18-m HiProt); 3 participants refused in-person visits due to COVID-19 concerns (1 per group), 1 participant moved out of state and only did a phone visit at follow-up (6-m HiProt), and 1 person had a hip replacement of the leg scanned at baseline (18-m HiProt)
Measure: Least Squares Mean (Standard Error); unit: cm^3
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt
Number analyzed (Participants) | 44 | 45 | 45
cm^3 | 0.72 (0.62) | 0.44 (0.64) | 1.11 (0.66)
Statistical Analysis 1: Comparison: RecProt vs 18-month HiProt; Test type: Superiority; p = 0.48, ANCOVA; Adjusted for age, sex, race
Statistical Analysis 2: Comparison: 6-month HiProt vs 18-month HiProt; Test type: Superiority; p = 0.22, ANCOVA; Adjusted for age, sex, race

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | RecProt | 6-month HiProt | 18-month HiProt
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 8/62 | 5/62 | 5/63
Other Adverse Events (participants affected / at risk) | 17/62 | 14/62 | 11/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RecProt (N=62) | 6-month HiProt (N=62) | 18-month HiProt (N=63)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cognitive Disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Knee Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Transurethral Resection Of Prostrate (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Shoulder Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Revision of Knee Replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hip Replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Umbilical Hernia Repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Reverse Shoulder Arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RecProt (N=62) | 6-month HiProt (N=62) | 18-month HiProt (N=63)
Sinusitis (Infections and infestations) | 7 (8) | 2 (2) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 7 (9) | 6 (6) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
We initially planned to end recruitment in August of 2020. However, our institution paused all in-person research from March 13, 2020 through May 31, 2020 due to the COVID19 pandemic. We extended our recruitment window through September 2020 but did not reach our target enrollment. The COVID19 pandemic also affected participant follow-up (a large number of out of window visits and a few who refused to return for in-person visits). The 6-month intervention also had to go remote for ~4 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT03074643/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT03074643/ICF_000.pdf